CLINICAL TRIAL: NCT06319313
Title: A Randomized, Controlled, Open-label Phase II/III Study of The Safety, Tolerability and Efficacy of JMT101 Combined With Docetaxel / HB1801 in Patients With sqNSCLC
Brief Title: Efficacy and Safety of JMT101 Combined Wth Docetaxel / HB1801 in Patients With Squamous Cell Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JMT101-013
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Squamous Cell Non-small Cell Lung Cancer
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JMT101+ docetaxel (Experimental)
  Interventions: Drug: JMT101; Drug: docetaxel
- JMT101+HB1801 (Experimental)
  Interventions: Drug: JMT101; Drug: HB1801
- HB1801 (Experimental)
  Interventions: Drug: HB1801

INTERVENTIONS:
Drug: JMT101 — JMT101, 6 mg/kg, IV infusion once every 2 weeks (one treatment cycle is 4 weeks). or 9 mg/kg, IV infusion once every 3 weeks.
  Arms: JMT101+ docetaxel; JMT101+HB1801
Drug: docetaxel — 50 mg/m2, IV infusion once every 2 weeks (one treatment cycle is 4 weeks). Or 75 mg/m2, IV infusion once every 3 weeks.
  Arms: JMT101+ docetaxel
Drug: HB1801 — 75 mg/m2, IV infusion once every 2 weeks (one treatment cycle is 4 weeks). Or 100 mg/m2, IV infusion once every 3 weeks.
  Arms: HB1801; JMT101+HB1801

SUMMARY:
This study is a phase II/III, randomized, controlled, open-label, multi-center study with safety run-in to evaluate the efficacy and safety of JMT101 combined with docetaxel/ HB1801 in Patients with Squamous cell non-small cell lung cancer （sqNSCLC）.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranged from 18 to 75 years old (inclusive), regardless of gender;
2. Pathological diagnosis as sqNSCLC, with EGFR highly expressed, without other driver genes
3. Tumor tissue available for central laboratory testing;
4. Disease progression after prior anti PD-1/PD-L1 and platinum containing chemotherapy
5. Measurable disease according to RECIST1.1;
6. Eastern Cooperative Oncology Group (ECOG) score 0-1 points;
7. Life expectancy ≥3 months
8. Adequate main organs and bone marrow function.
9. Patients must give informed consent to this study before the experiment and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Previously used anti EGFR, or docetaxel;
2. Central nervous system metastasis or meningeal metastasis;
3. Patients with high risk of bleeding due to tumor invasion of important arteries;
4. Uncontrolled or requiring repeated drainage of pleural effusion, pericardial effusion, or abdominal effusion;
5. The adverse reactions of previous anti-tumor treatments (including radiotherapy) have not yet recovered to CTCAE 5.0 evaluation ≤ level 1 except for toxicity such as alocepia or fatigue, which is judged to be of no safety risk by researchers;
6. Diagnosed as a second primary malignant tumor (except for skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder carcinoma, prostate carcinoma in situ, cervical carcinoma in situ and breast carcinoma in situ, etc.) within 5 years prior to the first administration of the study drug;
7. Have received anti-tumor treatments such as systemic chemotherapy, biological therapy, immunotherapy, radical radiotherapy chemotherapy, etc. within 28 days before the first dose of the study drug;
8. Have undergone major surgery (excluding needle biopsy) or suffered severe traumatic injury within 28 days before the first dose of study drug;
9. Have received a live viral vaccine or live-attenuated vaccine within 28 days before the first dose of study drug or plan to receive it during the study;
10. Have received palliative radiotherapy, small molecule targeted therapy, immunomodulatory drugs, NMPA approved modern traditional Chinese medicine preparations and other anti-tumor treatments, within 14 days before the first dose of study drug;
11. Those who use strong CYP3A4 inducers within 14 days before the first administration of the study drug, or those who use strong CYP3A4 inhibitors within 1 week, or those who cannot suspend the use of the above drugs during the study;
12. Have a history of serious cardiovascular disease;
13. Have a history of serious lung disease;
14. History of autoimmune diseases;
15. History of immunodeficiency
16. A history of gastrointestinal perforation and/or fistula within 6 months, or gastrointestinal obstruction and active inflammatory bowel disease within 28 days prior to the first study drug administration
17. Have infectious diseases requiring systemic anti-infective treatment;
18. Active hepatitis B; hepatitis C infection; syphilis infection, active tuberculosis;
19. Known hypersensitivity or intolerance to any component of EGFR monoclonal antibody, human serum albumin, docetaxel, and its excipients; Individuals known to be allergic and/or contraindicated to glucocorticoids
20. Women during lactation or pregnancy;
21. Any male and female patients with fertility who refuse to use effective contraceptive methods throughout the entire trial period and within six months after the last administration;
22. Other conditions that, in the opinion of the investigator, may affect the safety or compliance of drug treatment in this study, including but not limited to: psychiatric disorders, any severe or uncontrollable diseases, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 2 years
Overall Survival (OS) | Up to approximately 3 years
Incidence and severity of adverse events (AE) and serious adverse events (SAE) | Up to approximately 3 years
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 2 years
  PFS, defined as the time from randomization to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | Up to approximately 2 years
Duration of response（DOR） | Up to approximately 2 years
JMT101 Concentrations in Plasma | Up to approximately 2 years
Total and Free Docetaxel Concentrations in Plasma | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, M.D., Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No